CLINICAL TRIAL: NCT04729114
Title: Phase 1, Open-Label, Multicenter Study of Intramuscular PRL-02 Depot in Patients With Advanced Prostate Cancer
Brief Title: A Safety and Dose-finding Study of PRL-02 Depot in Men With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRL-02-1001
Record Dates: First submitted 2021-01-15; First posted 2021-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Metastatic Castration Resistant Prostate Cancer; Metastatic Castration-sensitive Prostate Cancer
Keywords: Testosterone; Testosterone suppression; metastatic castrate sensitive prostate cancer; metastatic castrate resistant prostate cancer; metastatic disease; prostate cancer; mCSPC; mCRPC; abiraterone; abiraterone decanoate; abiraterone acetate; Phase 1; Propella; ASP5541
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Prednisone; Dexamethasone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1a Dose Escalation: Group A (Experimental): Participants with metastatic castration-sensitive prostate cancer (mCSPC), nonmetastatic castration-sensitive prostate cancer (nmCSPC) with biochemical relapse, or metastatic castration-resistant prostate cancer (mCRPC) will receive escalating doses of PRL-02 + prednisone.
  Interventions: Drug: PRL-02 injection; Drug: prednisone
- Phase 1a Dose Escalation: Group B (Experimental): Participants with mCSPC, nmCSPC with biochemical relapse, or mCRPC will receive escalating doses of PRL-02 + dexamethasone.
  Interventions: Drug: PRL-02 injection; Drug: dexamethasone
- Phase 1a Dose Escalation: Group H (Experimental): Participants with mCSPC or mCRPC will receive escalating doses of PRL-02 + dexamethasone + enzalutamide.
  Interventions: Drug: PRL-02 injection; Drug: dexamethasone; Drug: enzalutamide
- Phase 1b Dose Expansion: Group D (Experimental): Participants with mCRPC with prior treatment with abiraterone acetate will receive escalating doses of PRL-02 + dexamethasone.
  Interventions: Drug: PRL-02 injection; Drug: dexamethasone
- Phase 1b Dose Expansion: Group E (Experimental): Participants with mCRPC with prior treatment with 1 of the following androgen receptor pathway inhibitor (ARPIs) (enzalutamide, apalutamide, and/or darolutamide) will receive escalating doses of PRL-02 + dexamethasone.
  Interventions: Drug: PRL-02 injection; Drug: dexamethasone

INTERVENTIONS:
Drug: PRL-02 injection — abiraterone decanoate for intramuscular injection
Drug: prednisone — Oral dose
  Arms: Phase 1a Dose Escalation: Group A
Drug: dexamethasone — Oral dose
  Arms: Phase 1a Dose Escalation: Group B; Phase 1a Dose Escalation: Group H; Phase 1b Dose Expansion: Group D; Phase 1b Dose Expansion: Group E
Drug: enzalutamide — Oral capsule
  Arms: Phase 1a Dose Escalation: Group H

SUMMARY:
Medicines that reduce the amount of testosterone in the body are commonly used to treat prostate cancer. PRL-02 depot is a potential treatment for men with advanced prostate cancer. It is given by an injection into the muscle. Men with advanced prostate cancer can take part in this study. Their cancer has come back after previous cancer treatment, or the previous cancer treatment they had didn't work.

The main aims of the study are:

* to check the safety of PRL-02 depot given with and without another medicine called enzalutamide.
* to check if the men can tolerate PRL-02 depot given with or without enzalutamide.
* to find a suitable dose of PRL-02 depot.

This study will be in 2 parts.

In the first part, different small groups of men will receive lower to higher doses of PRL-02 depot together with other medicines.

In the second part of the study, men who have previously taken a hormone therapy called abiraterone acetate or have previously taken 1 specific hormone therapy as part of their prostate cancer treatment can take part.

Men in both parts of the study will receive injections of PRL-02 depot into a muscle once every 12 weeks. They will also take dexamethasone or prednisone, or enzalutamide once a day. The other medicines they take depend on which group and which part of the study they are in.

During the study, the men will visit the clinic several times for health checks and scans.

After the final visit, men whose cancer has not become worse will continue to have health checks and scans every few months.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of adenocarcinoma of the prostate
* Phase 1a Dose Escalation Groups A and B: participants must have one of the following documented conditions:

  * mCSPC (must have documentation by positive bone scan [for bone disease] or metastatic lesions on computed tomography [CT] or magnetic resonance imaging [MRI] scan [for soft tissue])
  * nmCSPC with biochemical relapse of prostate cancer
  * mCSPC with oligometastatic prostate cancer (e.g., positron emission tomography positive)
  * mCRPC (must have documentation by positive bone scan [for bone disease] or metastatic lesions on CT or MRI scan [for soft tissue])
  * NOTE: For participants in the Dose Escalation Cohorts (including backfill) at each of the dose levels up to approximately 10 participants with ARPI-naïve mCRPC who have not received prior treatment with an ARPI (e.g., abiraterone acetate, enzalutamide, apalutamide, darolutamide) will be enrolled.
* Phase 1a Dose Escalation Groups A and B: participants with mCRPC must have evidence of disease progression defined as one or more of the following:

  * Evidence of radiographic progression of disease following the most recent prostate cancer treatment, defined as progressive disease on CT/MRI per RECIST v1.1 or on a bone scan per PCWG3.
  * PSA progression defined as the following:
* PSA nadir is defined as the lowest PSA during or after the most recent treatment. PSA progression is defined as an increased PSA of at least 25% and ≥1 ng/mL above the nadir confirmed by at least 2 measurements with a minimum of 1 week apart, and with at least 1 of the measurements within 90 days prior to screening.
* Participants with nmCSPC and biochemical recurrence, who had a radical prostatectomy (with or without radiotherapy) as the primary treatment for prostate cancer, must have a screening PSA ≥1 ng/mL. Participants with nmCSPC and biochemical recurrence who had radiotherapy only, as primary treatment for prostate cancer, must have a screening PSA ≥2 ng/mL above the nadir.
* Phase 1b Expansion Groups D and E: participants must have mCRPC Participants in Group D must have received prior treatment with abiraterone acetate, but must not have received treatment with other ARPIs (enzalutamide, apalutamide or darolutamide). Participants in Group E must have received prior treatment with only 1 of the following ARPIs: enzalutamide, apalutamide or darolutamide. Participants in both Groups D and E must have documented evidence of progression with one or more of the following:

  * Evidence of radiographic progression of disease following the most recent prostate cancer treatment, defined as progressive disease on CT/MRI per RECIST v1.1 or on a bone scan per PCWG3. Disease spread that is limited to the regional pelvic lymph nodes does not qualify as radiographic progression.
  * PSA progression defined as the following:
  * PSA nadir is defined as the lowest PSA during or after the most recent treatment. PSA progression is defined as an increased PSA of at least 25% and ≥1 ng/mL above the nadir confirmed by at least 2 measurements with a minimum of 1 week apart, and with at least 1 of the measurements within 90 days prior to screening.
* Participants with mCRPC must have undergone bilateral orchiectomy or received concurrent GnRH agonist or antagonist therapy for at least 6 weeks prior to the first dose of study drug.
* Participants with mCSPC or nmCSPC with biochemical recurrence should have received <6 months of ADT with a GnRH agonist or antagonist or have a history of bilateral orchiectomy (i.e., surgical or medical castration) within 6 months prior to Day 1. Castration therapy (i.e., medical or surgical) must have been started at least 14 days prior to Cycle 1 Day 1 and participants should have no radiographic evidence of disease progression or rising PSA levels after starting ADT and prior to Cycle 1 Day 1.
* A serum testosterone level <50 ng/dL at screening (for mCRPC participants only)
* Adequate muscle mass for an i.m. injection
* An ECOG PS of 0 or 1
* Adequate bone marrow reserve defined as:

  * Absolute neutrophil count (ANC) ≥1500/µL
  * Platelet count ≥100,000/µL
  * Hemoglobin ≥9 gm/dL
* Adequate renal function defined as a serum creatinine ≤1.5 × upper limit of normal (ULN) for the reference laboratory or a calculated creatinine clearance ≥50 mL/min as determined by a validated algorithm for calculating creatinine clearance
* Adequate hepatic function, defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN and total bilirubin ≤1.5 × ULN. Exception for elevated bilirubin secondary to Gilbert's disease. Confirmation of Gilbert's diagnosis requires: elevated unconjugated (indirect) bilirubin values; normal complete blood count in previous 12 months, blood smear, and reticulocyte count; normal aminotransferases and alkaline phosphatase in previous 12 months.
* Serum albumin ≥3 gm/dL and serum potassium ≥3.5 mEq/L
* Participants who are non-sterile and who are heterosexually active with a female partner of childbearing potential must be willing to use a highly effective means of contraception, such as a male condom plus spermicide, from the time of screening, throughout the total duration of the drug treatment, and until 12 weeks after the final dose of PRL-02 or enzalutamide (Group H).
* Participant is able to comply with study requirements throughout the study.

The Following Inclusion Criteria Apply to Dose Escalation Group H Only

* Participants must have one of the following documented conditions:

  * mCSPC (must have documentation of a positive PMSA-PET or positive bone scan [for bone disease] or metastatic lesions on CT or MRI scan [for soft tissue])
  * mCRPC (must have documentation of a positive PMSA-PET or positive bone scan [for bone disease] or metastatic lesions on CT or MRI scan [for soft tissue])
  * NOTE: For participants in the Dose Escalation Cohorts (including backfill) at each of the dose levels, the Sponsor may elect to enroll up to 10 participants with ARPI-naïve mCRPC who have not received prior treatment with an ARPI (e.g., abiraterone acetate, enzalutamide, apalutamide, darolutamide).
* Participants with mCRPC must have evidence of disease progression defined as one or more of the following:

  * Evidence of radiographic progression of disease following the most recent prostate cancer treatment, defined as progressive disease on CT/MRI per RECIST v1.1 or on a bone scan per PCWG3.
  * PSA progression defined as the following:
* PSA nadir is defined as the lowest PSA during or after the most recent treatment. PSA progression is defined as an increased PSA of at least 25% and ≥1 ng/mL above the nadir confirmed by at least 2 measurements with a minimum of 1 week apart, and with at least 1 of the measurements within 90 days prior to screening.
* Participant is able to swallow enzalutamide capsules whole.

Exclusion Criteria:

* Known active central nervous system (CNS) metastases. Note: Participants with CNS metastases that have been treated with surgery and/or radiation therapy, who are off pharmacologic doses of glucocorticoids, and who are neurologically stable are eligible.
* Impending bone fracture due to bone metastases
* Has a known additional malignancy beyond prostate cancer that required active treatment with the exception of any of the following:

  * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ carcinoma of any type
  * Adequately treated Stage I cancer from which the participant is currently in remission and has been in remission for ≥2 years
  * Any other cancer from which the participant has been disease-free for ≥5 years
* Clinically significant cardiac disease, defined as any of the following:

  * Clinically significant cardiac arrhythmias including bradyarrhythmia which are poorly controlled.
  * Congenital long QT syndrome
  * QT interval corrected by Fridericia's formula (QTcF) ≥450 msec at screening (based on average of triplicate ECGs at baseline). If the QT interval corrected for heart rate intervals (QTc) is prolonged in a participant with a pacemaker or bundle branch block, the participant may be enrolled in the study if confirmed by the Medical Monitor.
  * History of clinically significant cardiac disease or congestive heart failure greater than New York Heart Association (NYHA) Class II or left ventricular ejection fraction measurement of <50% at baseline. Participants must not have unstable angina (symptoms at rest) or new-onset angina within the last 3 months or myocardial infarction within the past 6 months [NYHA Classification 2014].
  * Uncontrolled hypertension, defined as systolic blood pressure (BP) >160 mmHg or diastolic BP >100 mmHg which has been confirmed by 2 successive measurements despite optimal medical management.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the 3 months before start of study medication (except for adequately treated catheter-related venous thrombosis occurring >1 month before the start of study medication).
* Received an investigational drug within 4 weeks or 5 half-lives (whichever is shorter) of the first dose of study drug.
* Received chemotherapy within 2 weeks or 5 half-lives (whichever is shorter) of the first dose of study drug.

  * Additional criteria: ARPI-naïve mCRPC participants enrolled in the Dose Escalation Cohorts (including backfill) must not have received prior chemotherapy in the mCRPC setting (prior receipt of chemotherapy in the mCSPC setting is allowed, if received at least 2 weeks or 5 half-lives prior to the first dose of study drug).
* Any unresolved NCI CTCAE criteria v5.0 Grade >2 toxicity from previous anticancer therapy at the Screening visit. Note: Participants receiving ongoing hormone replacement therapy for endocrine immune-related AEs without clinical symptoms will not be excluded.
* Has not recovered from recent major surgery or trauma
* Received a blood transfusion within 2 weeks of the first dose of study drug
* History of impaired pituitary or adrenal gland function (e.g., Addison's disease, Cushing's syndrome)
* Prior treatment with abiraterone acetate, orteronel. Exception: participants in Phase 1b Expansion Group D will have received prior abiraterone acetate, and participants in Group H may have received prior treatment with abiraterone acetate.
* Current treatment with systemic ketoconazole or any other CYP17 inhibitor. Participants who have received systemic ketoconazole or any other CYP17 inhibitor must have discontinued these agents ≥4 weeks prior to the first dose of study drug.
* Prior systemic treatment with an azole drug (e.g., fluconazole, itraconazole) within 4 weeks of first dose of study drug.
* Prior treatment with estrogens within 12 weeks of the first dose of study drug
* Need for systemic glucocorticoids greater than replacement doses; the use of topical, intraocular, inhalational, intranasal, or intra-articular glucocorticoids is permitted.
* Prior use of any herbal products that could decrease PSA levels (e.g., saw palmetto) within 4 weeks of the first dose of study drug. Participants must agree not to use such herbal products during study participation.
* Use of biotin (i.e., vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg [NIH-ODS 2022]. Note: Participants who switch from a high dose to a dose of 30 µg/day or less prior to first dose of study drug are eligible for study entry.
* Required concomitant use of strong inducers of CYP3A4, except for enzalutamide given as study drug in Group H
* Known hypersensitivity to PRL-02, abiraterone, abiraterone decanoate, prednisone, or dexamethasone or any of their excipients or components.
* Has jaundice or known current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M [IgM] positive), hepatitis B (hepatitis B virus surface antigen [HBsAg] positive, confirmed by polymerase chain reaction [PCR]), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid)
* Hemoglobin A1c (HbA1c) >10% in participants previously diagnosed with diabetes mellitus. HbA1c >8% in participants whose diabetes mellitus is previously undiagnosed. (Excluded participants may be rescreened after referral and evidence of improved control of their condition).
* Uncontrolled infection with human immunodeficiency virus (HIV)+. Exception: participants with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible.
* Body mass index >40 kg/m2

The Following Exclusion Criteria Apply to Dose Escalation Group H Only

* Clinically significant cardiac disease, defined as any of the following:

  * NYHA class III or IV congestive heart failure or a history of NYHA class III or IV congestive heart failure, unless a screening echocardiogram or multigated acquisition scan performed within 3 months before the randomization date demonstrates a left ventricular ejection fraction of ≥45%
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
  * Hypotension as indicated by systolic BP <86 mm Hg at screening
  * Bradycardia as indicated by a heart rate of ≤45 beats per minute on the screening ECG
* Participant has a history of seizure or any condition that may predispose to seizure.
* Use or required use of any prohibited medication.
* Participant has a gastrointestinal disorder affecting absorption.
* Participant has shown hypersensitivity reaction to the active pharmaceutical ingredient or any of the study capsule components, including Labrasol®, butylated hydroxyanisole, and butylated hydroxytoluene.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  A DLT is defined as any event meeting the DLT criteria during the first 28 days of each Dose Escalation treatment regardless of attribution to the study drug unless due to underlying disease or extraneous causes.
Number of Participants with Adverse Events (AEs) | Up to 4 years
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Number of Participants with Serious Adverse Events (SAEs) | Up to 4 years
  An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important events.
Number of Participants with laboratory value abnormalities and/or AEs | Up to 4 years
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 4 years
  Number of participants with potentially clinically significant ECG values.
Number of Participants with vital sign abnormalities and/or AEs | Up to 4 years
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with physical exam abnormalities and/or AEs | Up to 4 years
  Number of participants with potentially clinically significant physical exam values or symptoms.
Number of Participants with Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 4 years
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Testosterone Suppression of Participants as Assessed by Testosterone Levels | Up to 4 years
  Reduction in testosterone will be summarized by group and dose level.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of Abiraterone in plasma: Maximum Concentration (Cmax) | Up to 455 days
  Cmax will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: Cmax | Up to 455 days
  Cmax will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: Cmax | Up to 455 days
  Cmax will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: Minimum Concentration (Cmin) | Up to 455 days
  Cmin will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: Cmin | Up to 455 days
  Cmin will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: Cmin | Up to 455 days
  Cmin will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: Time of maximum concentration (tmax) | Up to 455 days
  tmax will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: tmax | Up to 455 days
  tmax will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: tmax | Up to 455 days
  tmax will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: apparent volume of distribution (Vd/F) | Up to 455 days
  Vd/F will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: Vd/F | Up to 455 days
  Vd/F will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: Vd/F | Up to 455 days
  Vd/F will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: oral clearance (CL/F) | Up to 455 days
  CL/F will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: CL/F | Up to 455 days
  CL/F will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: CL/F | Up to 455 days
  CL/F will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: area under the curve from time 0 to the time of the last measurable concentration (AUClast) | Up to 455 days
  AUClast will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: AUClast | Up to 455 days
  AUClast will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: AUClast | Up to 455 days
  AUClast will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: Area Under the Concentration-time Curve from the Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 455 days
  AUCinf will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: AUCinf | Up to 455 days
  AUCinf will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: AUCinf | Up to 455 days
  AUCinf will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: area under the plasma concentration-time curve during a dosage interval (AUCtau) | Up to 455 days
  AUCtau will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: AUCtau | Up to 455 days
  AUCtau will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: AUCtau | Up to 455 days
  AUCtau will be recorded from the PK plasma samples collected.
PK of Abiraterone in plasma: Terminal Elimination Half-life (t1/2) | Up to 455 days
  t1/2 will be recorded from the PK plasma samples collected.
PK of Abiraterone Decanoate in plasma: t1/2 | Up to 455 days
  t1/2 will be recorded from the PK plasma samples collected.
PK of Abiraterone Metabolite in plasma: t1/2 | Up to 455 days
  t1/2 will be recorded from the PK plasma samples collected.
Composite Response Rate | Up to 4 years
  Composite responses will be defined as meeting any one of the following criteria:
  Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 with a minimum interval for confirmation of complete response (CR) or partial response (PR) of 4 weeks or; prostate specific antigen (PSA) decline of ≥50% confirmed by a second consecutive PSA assessment at least 3 weeks later, or;
  Conversion of circulating tumor cell (CTC) count to <5 cells/7.5 mL blood nadir confirmed by an additional assessment at least 3 weeks later (for participants with a CTC count of ≥5 cells/7.5 mL blood at screening).
Best overall response (BOR) per RECIST v1.1 | Up to 4 years
PSA decline of ≥50% response from baseline (PSA50) | Up to 4 years
  Defined as ≥50% decline in PSA from baseline, confirmed by a second consecutive PSA assessment at least 3 weeks later.
PSA decline of ≥90% response from baseline (PSA90) | Up to 4 years
  Defined as ≥90% decline in PSA from baseline, confirmed by a second consecutive PSA assessment at least 3 weeks later.
Percentage of participants achieving a PSA level <0.2 ng/mL | Up to 4 years
Duration of response (DOR) | Up to 4 years
  DOR is defined as the length of time from date of first documented response using CTC count and/or PSA and/or RECIST v1.1 and Prostate Cancer Working Group 3 (PCWG3) until date of documented progression or death from any cause.
Radiographic progression-free survival (rPFS) | Up to 4 years
  rPFS is defined as the time from first dose of study drug to documented progression or death using RECIST v1.1 or PCWG3.
Overall response rate (ORR) using RECIST v1.1 | Up to 4 years
  ORR is defined as percentage of patients with measurable disease at baseline who achieved a complete or partial response in their soft tissue disease using the RECIST v1.1 criteria.
Time to PSA progression | Up to 4 years
  The time from first dose of study drug to documented PSA progression.
Overall survival (OS) | Up to 4 years
  OS is defined as the time from the first dose of study drug to the date of death due to any cause.
Time to first symptomatic skeletal-related event (SSRE) | Up to 4 years
  The time from first dose of study drug to first documented symptomatic skeletal-related event: Use of radiation therapy to prevent or relieve skeletal symptoms, occurrence of new symptomatic pathologic bone fractures (vertebral or nonvertebral) with radiologic documentation, occurrence of spinal cord compression with radiologic documentation, orthopedic surgical intervention for bone metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development, Inc.
Locations (25):
- United States (24):
  - Arizona Urology Specialists, Tucson, Arizona
  - Los Angeles Cancer Network, Anaheim, California
  - Providence Medical Group Oncology Santa Rosa, Santa Rosa, California
  - Florida Urology Partners, Tampa, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - First Urology, Jeffersonville, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - National Cancer Institute, Bethesda, Maryland
  - Chesapeake Urology, Towson, Maryland
  - XCancer Center Omaha/Urology Cancer Center, Omaha, Nebraska
  - Garden Sate Urology, Morristown, New Jersey
  - New Mexico Oncology Hematology Consultants Ltd, Albuquerque, New Mexico
  - Duke Cancer Center, Durham, North Carolina
  - Helios Clinical Research, LLC, Middleburg Heights, Ohio
  - Toledo Clinical Cancer Center, Toledo, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates PC, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
- Pan American Center for Oncology Trials, LLC, San Juan, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/